CLINICAL TRIAL: NCT03424148
Title: Open-label, Prospective, Multicenter Study to Evaluate the Cutera Excel V™ Laser and a Micro-Lens Array Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-17-EV11
Record Dates: First submitted 2018-01-24; First posted 2018-02-06 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Scarring; Skin Aging
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Excel V™ Laser & Micro-Lens Array Attachment (Other): Treatment with Excel V™ Laser and a Micro-Lens Array Attachment for skin quality
  Interventions: Device: Excel V™ Laser & Micro-Lens Array Attach

INTERVENTIONS:
Device: Excel V™ Laser & Micro-Lens Array Attach — Subjects will receive laser treatments

SUMMARY:
Open-label, Prospective, Study to Evaluate the Cutera excel V laser at 532 nm in a low fluence, high repetition rate mode and the Micro-Lens Array attachment used with excel V laser at 1064 nm and 532 nm for the improvement of skin quality.

DETAILED DESCRIPTION:
This is an open-label, prospective, study in approximately 60 male or female subjects, age 18 to 65 years who desire laser treatment for the improvement of rhytides, lentigines, pigmentation, erythema, telangiectasia, pore size and skin texture. Subjects may undergo a 2mm punch biopsy a treatment area up to 72 hours post treatment and at a designated follow-up period per Investigator discretion. Subjects will receive laser treatments. Subjects will return to the site after final study treatment for two follow-up visits: 6 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to read, understand and sign the Informed Consent Form.
2. Female or Male, 18 to 65 years of age (inclusive).
3. Fitzpatrick Skin Type I - VI.
4. Must be willing to have Cutera excel V laser treatments and able to adhere to the treatments, follow-up visit schedule, and post-treatment care instructions.
5. Willing to have very limited sun exposure and use sunscreen on the treatment area every day for the duration of the study, including the follow-up period.
6. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation (educational and/or marketing), publications, and any additional marketing purposes.
7. Agree to not undergo any other cosmetic procedure(s) or treatment(s) on the face during the study and has no intention of having such procedures performed during the course of the study.
8. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.,

Exclusion Criteria:

1. Participation in a clinical trial of another drug, or device administered to the treatment area, within 3 months prior to enrollment or during the study.
2. Any type of prior cosmetic treatment to the target area within 6 months of study participation, such as laser procedures, facial fillers, toxins and those used for general aesthetic correction.
3. Use of prescription topicals in the treatment area within one month prior to treatment or use of topical agents one week prior to treatment that may cause facial sensitivity.
4. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including but not limited to, open lacerations or abrasions, hidradenitis, rash, infection , or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion).
5. Pregnant and/or breastfeeding, or planning to become pregnant.
6. Significant concurrent illness, such as diabetes mellitus, immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or using immunosuppressive medication.
7. Hypersensitivity to light exposure.
8. Any use of medication that is known to increase sensitivity to light according to the Investigator's discretion.
9. History of keloid scarring, hypertrophic scarring or abnormal wound healing or prone to bruising.
10. Has a history of squamous cell carcinoma or melanoma in the treatment area.
11. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders.
12. A history or active skin condition that in the opinion of the Investigator may interfere/confound with the treatment.
13. History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
14. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
15. History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation, or any that are considered not acceptable by the study investigator.
16. Has used oral isotretinoin (Accutane or therapeutic vitamin A supplements of ≥ 10,000 units per day) within 12 months of initial treatment or plans on using during the course of the study (note: skin must regain its normal degree of moisture prior to treatment, e.g. lack of noticeable skin flaking and peeling).
17. Excessively tanned or active sun tan in facial area to be treated, or unable/unlikely to refrain from tanning during the study.
18. Excessive facial hair in the area to be treated (beards, sideburns, and/or moustache,) that would interfere with diagnosis, assessment, and treatment.
19. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study, including excessive alcohol or drug abuses, or a condition that would compromise the subject's ability to comply with the study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cutera Research Center, Brisbane, California
  - Center for Dermatology and Laser Surgery, Sacramento, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Excel V™ Laser & Micro-Lens Array Attachment: Treatment with Excel V™ Laser and a Micro-Lens Array Attachment
Period: Overall Study
Arm/Group | Excel V™ Laser & Micro-Lens Array Attachment
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Excel V™ Laser & Micro-Lens Array Attachment
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Study Effectiveness for Skin Aesthetic Improvement
Description: Efficacy of treatment(s) with Cutera excel V™ laser and the Micro-Lens Array attachment as assessed by the study investigator using GAIS: Global Aesthetic Improvement Scale Higher scores indicate better outcomes (+4=Very Significant Improvement, +3=Significant Improvement, +2=Moderate Improvement, +1=Mild Improvement, or 0=No Change) Subjects had one assessment done at either the 6 or 12 week follow up, and GAIS values from the 6 and 12 week follow up visits were summed together to calculate the mean
Time Frame: 6 or 12 weeks after the final treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Excel V™ Laser & Micro-Lens Array Attachment
Number analyzed (Participants) | 8
score on a scale | 1.25 (0.71)

ADVERSE EVENTS:
Time Frame: 12 weeks post final treatment, up to 9 months
Arm/Group | Excel V™ Laser & Micro-Lens Array Attachment
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Excel V™ Laser & Micro-Lens Array Attachment (N=10)
Erythema (Skin and subcutaneous tissue disorders) | 10
Edema (Skin and subcutaneous tissue disorders) | 9
Purpura (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT03424148/Prot_SAP_000.pdf